CLINICAL TRIAL: NCT06619639
Title: Cluster Randomized Trial of a Novel Social-emotional Learning Curriculum in an After-school Program for Youth, 11-14 Years
Brief Title: Feasibility of a Social-emotional Learning Curriculum in an After-school Program for Youth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Brendan Andrade, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/111; Les Lois Shaw Foundation (Other: Les Lois Shaw Foundation)
Record Dates: First submitted 2024-09-17; First posted 2024-10-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Feasibility Studies; Efficacy of Intervention; Social Emotional Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual programming control (implement beyond 3:30 programming as usual) (No Intervention): Groups assigned to the usual programming control arm will deliver regular beyond 3:30 programming.
- Social-emotional learning curriculum (Experimental): The intervention is the EMPOWER social-emotional learning curriculum.
  Interventions: Behavioral: Social-emotional learning curriculum

INTERVENTIONS:
Behavioral: Social-emotional learning curriculum — EMPOWER is a 16-week social-emotional learning curriculum that is integrated into the after-school program context.
  Arms: Social-emotional learning curriculum

SUMMARY:
The goal of this cluster randomized trial is to:

1. primary purpose: to determine the feasibility of a novel social-emotional learning curriculum when implemented in the beyond 3:30 after school program; 2a. secondary purpose: to determine whether the novel social-emotional learning curriculum has positive effects youth social emotional learning skills; 2b. secondary purpose: to determine whether the novel social-emotional learning curriculum has positive effects on youth resilience and overall functioning.

Participants:

1. Beyond 3:30 facilitators
2. Youth aged 11-14 who participate in the beyond 3:30 program
3. Parents of youth who participate in the beyond 3:30 program

The main questions this study aims to answer are:

Primary Objectives:

1. Is the novel social-emotional curriculum feasible within the beyond 3:30 after school program?
2. Is the novel social-emotional curriculum acceptable within the beyond 3:30 after school program?
3. Is the novel social-emotional curriculum appropriate within the beyond 3:30 after school program?

Secondary Objectives: Social-emotional learning skills 1. Have youth social-emotional learning skills improved as a result of participating in the novel social-emotional learning curriculum?

Secondary Objectives: Resilience and overall functioning

1. Have youth resilience abilities and overall functioning improved as a result of participating in the novel social-emotional learning program?

   Comparator:

   Primary objective: Feasibility - There is no comparison group for the feasibility objectives.

   Secondary objective: Social-emotional learning skills
   * The investigators will compare the intervention arm [10 sites within the beyond 3:30 program who will implement the EMPOWER social-emotional learning curriculum] with the usual programming control arm [10 sites within the beyond 3:30 program who will implement the usual beyond 3:30 program]

   Secondary objective: Resilience and overall functioning

   - The investigators will compare the intervention arm [10 sites within the beyond 3:30 program who will implement the EMPOWER social-emotional learning curriculum] with the usual programming control arm [10 sites within the beyond 3:30 program who will implement the usual beyond 3:30 program]

   Measures:

   Primary Objective: Feasibility

   After school program staff participants in the intervention arm will be asked to complete:

   - 3 feasibility measures (feasibility, acceptability, appropriateness of intervention) every 4-weeks after each social-emotional module they complete teaching.

   - weekly fidelity checklists to assess feasibility.

   Youth participants in the intervention arm will be asked to complete:

   - the intervention appropriateness measure during the post-curriculum data collection time point.

   Secondary Objective: Social-emotional learning skills

   After school program staff participants in both intervention and usual programming arms will be asked to complete the following measure pre- and post-curriculum implementation:

   - social-emotional learning skills measure for each youth aged 11-14 years in their class.

   Youth participants in both intervention and usual programming arms will be asked to complete the following measure pre- and post-curriculum implementation:

   - social-emotional learning skills measure Parents participants whose youth are in the intervention arm will be asked to participate in an interview.

   Secondary objective: Resilience and overall functioning

   After school program staff participants in both intervention and usual programming arms will be asked to complete the follow measures pre- and post-curriculum implementation:

   - overall functioning measure for each youth aged 11-14 years in their class.

   Youth participants in both intervention and usual programming arms will be asked to complete:
   * resilience measure

DETAILED DESCRIPTION:
The EMPOWER project is a community-academic partnership between 2 after school programs (beyond 3:30 and Visions of Science) and a mental health teaching hospital (Centre for Addiction and Mental Health). The main objective of this project is to bolster youth mental well-being by developing a novel social-emotional learning curriculum that after school programs can embed into their existing activities.

The curriculum is designed to improve youth's social emotional learning skills through the integration of short social-emotional learning lessons that are embedded into existing programming within an after school program. The curriculum is based on the Collaborative for Academic, Social and Emotional Learning's five core SEL competencies that include self-awareness, self-management, social awareness, relationship skills and decision-making.

The investigators have designed a pilot study to test the feasibility and efficacy of the EMPOWER social-emotional learning curriculum. Beyond 3:30 has 20 sites that are housed in schools across socially and economically vulnerable locations. We will randomize (based on class size and sites who participated in a previous trial of a part of the curriculum) 10 sites to be in the intervention and 10 sites to be in the usual programming control. The intervention arm will implement the 16-week EMPOWER social-emotional learning curriculum, while the usual programming control arm will implement regular beyond 3:30 programming.

ELIGIBILITY:
INCLUSION:

Youth participants must meet the following inclusion criteria:

1. Must be a youth aged 11-14 years attending the beyond 3:30 program
2. Must sign and date the informed consent form
3. Must speak and understand English

Staff participants must meet the following inclusion criteria:

1. Must be a facilitator of the beyond 3:30 program
2. Must sign and date the informed consent form
3. Must speak and understand English

Caregiver/parent participants must meet the following inclusion criteria:

1. Must be a caregiver/parent of a youth aged 11-14 years attending the beyond 3:30 program. Caregivers/parents whose children decide not to participate in data collection are still able to participate in an interview post-SEL curriculum implementation.
2. Must sign and date the informed consent form
3. Must speak and understand English

EXCLUSION; None

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 20-weeks
  Staff in the active intervention arm will complete the Feasibility of Intervention (Weiner et al., 2017) measure after each social-emotional domain (self-awareness, self-management, social awareness and relationship skills, decision-making) is taught. This is a 4-item, 5-point Likert-type scale that measures a composite feasibility of intervention score.
Acceptability of Intervention | 20-weeks
  Staff in the active intervention arm will complete the Acceptability of Intervention Measure (Weiner et al., 2017) measure after each social-emotional domain (self-awareness, self-management, social awareness and relationship skills, decision-making) is taught. This is a 4-item, 5-point Likert-type scale that measures a composite acceptability of intervention score.
Intervention Appropriateness | 20-weeks
  Staff in the active intervention arm will complete the Intervention Appropriateness (Weiner et al., 2017) measure after each social-emotional domain (self-awareness, self-management, social awareness and relationship skills, decision-making) is taught. This is a 4-item, 5-point Likert-type scale that measures a composite appropriateness of intervention scale. Youth in the intervention arm will complete the intervention appropriateness (Weiner et al., 2017) scale post-SEL curriculum implementation.

SECONDARY OUTCOMES:
Overall functioning | 20 weeks
  KIDSCREEN 10 (Child Public Health, 2023) is a 10-item, 5-point Likert-type scale that measures global quality of life.
  * Staff in active intervention and usual programming arms will complete an adapted version of the KIDSCREEN for each youth they work with (avg. 20 youth/site) pre- and post-EMPOWER SEL curriculum intervention.
  * Youth in active intervention and usual programming arms will complete the KIDSCREEN pre- and post-EMPOWER SEL curriculum intervention.
Resilience | 20 weeks
  Connor-Davidson Resilience Scale (CD-RISC-10; 2007) is a 10-item, 5-point Likert-type scale that measures overall resilience.
  - Youth in active intervention and usual programming arms will complete this measure pre- and post-EMPOWER SEL curriculum intervention.
Social-emotional learning skills | 20 weeks
  Social Skills Improvement System - Social Emotional Learning (SSIS-SEL Brief Scale; (Elliot et al., 2020) is a 20-item, 4-point Likert-type scale that measures self-awareness, self-management, social awareness, relationship skills, and decision making as a composite score of social-emotional competency.
  * Staff in both active intervention and usual programming arms will complete the SSIS-SEL Brief Scale for each youth they work with (avg. 20 youth/site) pre- and post-EMPOWER SEL curriculum intervention.
  * Youth in active intervention and usual programming arms will complete the SSIS-SEL Brief Scale pre- and post-EMPOWER SEL curriculum intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan F Andrade, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balter AS, Racine N, Al-Khooly D, Somir I, Bandoles E, Utchay C, Sylvestre D, Sibalis A, Suri A, Pierre S, Parkes S, Quesnelle S, Brodkin S, Andrade BF. Strengthening Youth Emotional and Behavioral Well-Being Through Community-Academic Partnership: The EMPOWER Project. Health Promot Pract. 2025 Sep;26(5):837-840. doi: 10.1177/15248399241255372. Epub 2024 Jul 27. PMID 39066621